CLINICAL TRIAL: NCT01596543
Title: Thr Effect of Partial and Complete Sleep Deprivation on Heat Tolerance
Brief Title: The Effect of Partial and Complete Sleep Deprivation on Heat Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: International Diabetes Federation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-11-8728-AD-CTIL
Record Dates: First submitted 2012-05-06; First posted 2012-05-11 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Sleep Deprivation
Keywords: sleep; HTT; heat illness
MeSH Terms: conditions — Sleep Deprivation; Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sleep deprivation (Experimental): The research contains only one arm. The subjects will be tested with no sleep deprivation (which will be used as a control measurement) and with partial and complete sleep deprivation.
  Interventions: Other: partial and complete sleep deprivation

INTERVENTIONS:
Other: partial and complete sleep deprivation — The subjects will visit our labs 4 times. The second visit will be used as the experimental control. During the third and fourth visits the subject will go through an exercise heat tolerance test and a measurement of their physiological efficiency after a partial and complete sleep deprivation, respectively.

SUMMARY:
The purpose of the present study is to evaluate the effect of partial and complete sleep deprivation on exercise heat tolerance. Twelve healthy young male volunteers will participate in the study. They will arrive to our lab four times, in each visit the will undergo VO2 test and Heat Tolerance Test (HTT) after sleeping different amount of hours.

DETAILED DESCRIPTION:
The volunteers will arrive to our lab fout times- During their first visit they will go through a VO2 max test in order to evaluate their aerobic fitness, and their physiological efficiency will be measured. During their second visit they will go through an exercise heat tolerance test according to our validated protocol after a full night sleep. During the third and fourth visit they will go through an exercise heat tolerance test and a measurement of their physiological efficiency after a partial and complete sleep deprivation, respectively. The physiological tests will take place in the heat chamber that is located at the Heller Institute of Medical Research. The results will be then analyzed, and a comparison between the physiological measurements during the heat tolerance tests and the physiological efficiency tests after the various sleep conditions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* healthy
* after medical checkup
* after signing concent form

Exclusion Criteria:

* heart disease
* respiratory disease
* baseline bp above 140/90 mmHg
* sleep disorders
* diabetes
* anhydrosis
* skin disease
* acute illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
oxygen consumption | experimental days 1,3,4
  volunteer's oxygen consumption (VO2) will be monitored continuously with a metabolic chart (ZAN), while running for 10 min on a treadmill under comfortable environmental conditions.Each volunteer will undergo the test 4 times.

SECONDARY OUTCOMES:
Skin temperature | experimental days 2,3,4
  The volunteers will undergo Heat Tolerance Test (HTT). Their skin temperature will be measured by skin thermistors and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Rectal temperature | experimental days 2,3,4
  The volunteers will undergo heat tolerance test. Their rectal temperature will be measured by rectal thermistor and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Heart rate | experimental days 1,2,3,4
  During the HTT (Heat Tolerance Test) and the VO2 test heart rates will be monitored continuously and will be stored by a heart rate wristwatch, (POLAR, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Druyan, M.D, Principal Investigator — The Institute of Military Physiology
Locations (1):
- Heller Institute of Medical Research, Tel-Hashomer, Ramat-Gan, Israel

REFERENCES:
- [Derived] Muginshtein-Simkovitch E, Dagan Y, Cohen-Zion M, Waissengrin B, Ketko I, Heled Y. Heat tolerance after total and partial acute sleep deprivation. Chronobiol Int. 2015 Jun;32(5):717-24. doi: 10.3109/07420528.2015.1030409. Epub 2015 May 8. PMID 25955404